CLINICAL TRIAL: NCT04926350
Title: Resistance Exercise Breaks Improve Ratings of Discomfort and Fatigue in College
Brief Title: Resistance Exercise Breaks Improve Ratings of Discomfort and Fatigue in College Students (REX)
Acronym: REX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University Kingsville (Other)
Responsible Party: Principal Investigator, Robert J. Kowalsky, Assistant Professor, Texas A&M University Kingsville
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 12183 / 2018-018-A1-R1
Record Dates: First submitted 2021-06-02; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Sedentary Behavior; Fatigue; Sleepiness; Pain
Keywords: physical activity; resistance exercise
MeSH Terms: conditions — Sedentary Behavior; Fatigue; Sleepiness; Pain; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Tracking of outcomes during a normal week
- Resistance Exercise (Experimental): Tracking of outcomes during a normal week with the addition of daily resistance exercise breaks (8 breaks per day)
  Interventions: Behavioral: Resistance Exercise

INTERVENTIONS:
Behavioral: Resistance Exercise — 8 total resistance exercises that target all major muscle groups
  Arms: Resistance Exercise

SUMMARY:
The purpose of this investigation is to determine the impact of simple resistance exercise breaks on physical activity and prolonged sedentary behavior as well as on ratings of discomfort, fatigue, and sleepiness. Participants will be enrolled in a cross-over designed study, where they will be assessed for normal activity patterns and ratings of discomfort, fatigue, and sleepiness during a typical week and compared to a week where they engage in hourly resistance exercise breaks. Subjects will also complete a feasibility questionnaire at the end to determine if such programming could be implemented into daily living. The hypothesis is that engaging in these simple, hourly resistance breaks will result in decreased ratings of discomfort, fatigue, and sleepiness as well as ratings of high feasibility for implementation of similar resistance exercise programming into their normal, everyday life. Total time spent enrolled in the study will be 4 weeks, however, the participants will only need to report to the lab on 5 different occasions totaling 120 minutes split over those 5 days. Visit one will be roughly 60 minutes long, with the following 4 visits taking roughly 15 minutes each with a visit at the beginning of the week and end of the week for both the control and experimental week.

DETAILED DESCRIPTION:
Each participant will encounter 1 familiarization session and 4 other brief sessions throughout the study. The study will consist of a 4 week protocol, with the first week having one familiarization visit, the second week being a baseline assessment week of normal activity, the third week being a washout period where no assessment is being done, and the fourth week being another assessment week while also completing the hourly resistance exercise breaks. Total time required for participants to report to the laboratory will be 120 minutes, but will be split over 5 visits (visit one: 60 minutes, visit two: 15 minutes, visit three: 15 minutes, visit four: 15 minutes, visit 5: 15 minutes).

The familiarization day will consist of the subject going through an initial screening to determine eligibility to participate in the study, as well as signing the informed consent. Following this, the participants will complete questionnaires to assess characteristics of interest (age, ethnicity, and activity level) and any other relevant characteristics deemed to be important to describe the population. Individuals will then be shown the journals and how to use them (journal attached). These journals will be used to track their ratings of discomfort, fatigue, and sleepiness across each of the days for both assessment weeks. Next, the individual will be shown each of the exercises that will be used during the resistance exercise break week and will be asked by the PI to complete each one so that the PI can provide any feedback to correct the movements to ensure safety. The subjects will also be given typed handouts describing each exercise in detail for their own records. Lastly, the subjects will be shown the activity monitors and how they will be applied to their body and how to replace the adhesive tape if needed during the weeks they are wearing the device (See attachment). This visit is expected to last roughly 60 minutes.

Visit #2 (week 2) will take place Monday morning at 8:00 am the week following the familiarization visit and will last roughly 15 minutes. At this visit, the PI will secure the activity monitor to the subject, and provide extra adhesive strips if needed. The subject will also receive their journal for the week to assess discomfort, fatigue, and sleepiness. The subject will be asked to track their ratings at three separate time points (morning: between 8:00-9:00 am, mid-day: between 1:00-2:00 pm, and evening: between 6:00-7:00 pm) across each of the next 7 days (Monday-Sunday). During the 7 days, the subject will be wearing the activity monitor the entire time (awake and sleep) and will only be removed if swimming/bathing (shower is ok: waterproof). The subject will be asked to go about their week as they normally do, with no extra intervention, to track activity and ratings for a typical week. This week will not have them completing any exercises and will serve as a control week for assessing physical activity pattern. Total time spent filling out the journal will be roughly 2-3 minutes per time, so roughly 9 minutes per day, and 63 minutes for the entire week.

Visit #3 (week 3) will take place on the Monday following the 7 days of assessment. The PI will remove the activity monitor and collect any extra adhesive strips. The subject will also turn in their journal that was used to track their ratings for the previous week. This visit will take roughly 15 minutes. At this point the subject will be allowed to leave and begin the washout week with no assessment.

Visit #4 (Week 4) will take place Monday morning at 8:00 am the week following the washout week and will last roughly 15 minutes. At this visit, the PI will secure the activity monitor to the subject, and provide extra adhesive strips if needed. The subject will also receive their journal for the week to assess discomfort, fatigue, and sleepiness. The subject will be asked to track their ratings at three separate time points (morning: between 8:00-9:00 am, mid-day: between 1:00-2:00 pm, and evening: between 6:00-7:00 pm) across each of the next 7 days (Monday-Sunday). During the 7 days, the subject will be wearing the activity monitor the entire time (awake and sleep) and will only be removed if swimming/bathing (shower is ok: waterproof). The subject will also now be asked to completely hourly resistance exercise breaks each hour for a total of eight exercises per day. Subjects will be asked to complete 2 sets of 15 repetitions each for all eight exercises with a minute rest in between sets. Each break should take less than 5 minutes. All exercises will be low intensity that utilize their own body weight as resistance or use a light resistance band with handles. Exercises will be split in groups of 4 with one group in the morning and one in the afternoon, with one exercise taking place per time slot. Time slots will be as follows: between 9:00-10:00 am, 10-11:00 am, 11:00-12:00 pm, and 12:00-1:00 pm, as well as from 2:00-3:00 pm, 3:00-4:00 pm, 4:00-5:00pm, and 5:00-6:00pm. Each exercise in detail is described in the handout that will be given to each participant (attached). This will require the participant to be engaged in exercise roughly 24 minutes per day, for a total of 168 minutes of exercise for the week. The participant will also be filling out the journals for the second assessment week similar to the first assessment week, totaling roughly 63 minutes for the week completing the journals.

Visit #5 (week 4) will take place on the Monday following the second week of 7 day assessments. The PI will remove the activity monitor and collect any extra adhesive strips. The subject will also turn in their journal that was used to track their ratings for the previous week. Finally the subjects will be asked to complete a brief questionnaire about the feasibility of such programming in their daily life. This visit will take roughly 15 minutes. This will complete the subject's participation in the study.

Information about participants and related to this study will be kept confidential to the extent permitted or required by law. Hard copies of the data collection materials will kept under lock and key for a period of no less than five years, then disposed of as sensitive materials according to University policy/procedures. Data collections sheets and informed consent documents will be stored separately. All data collection forms will not have any identifiable information on them and will have an ID number to link the information to the participant. Form linking participant name to ID will be kept electronically in a password protected computer file along with the reduced and analyzed data that is collected.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, participants need to be actively taking college classes, between the ages of 18 and 35 years old, and have no contraindications to participating in physical activity.

Exclusion Criteria:

* Any contraindication for physical activity participation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Physical activity | a week
  number of daily steps taken
Sedentary behavior | a week
  amount of daily sedentary behavior accumulated

SECONDARY OUTCOMES:
Physical discomfort | assessed morning, mid-day, and evening over a week period
  Subjective ratings of discomfort for 15 separate sites on the body using 100 pt visual analog scale
Physical Fatigue | assessed morning, mid-day, and evening over a week period
  Subjective rating of physical fatigue using a single 100 pt visual analog scale
Mental Fatigue | assessed morning, mid-day, and evening over a week period
  Subjective rating of mental fatigue using a single 100 pt visual analog scale
Sleepiness | assessed morning, mid-day, and evening over a week period
  Single value reported from Karolinska sleeping scale ranging from 1 to 9

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kowalsky, Ph.D., Principal Investigator — Texas A&M University Kingsville
Locations (1):
- Texas A&M University-Kingsville Human Performance Laboratory, Kingsville, Texas, United States

IPD SHARING:
Plan to Share IPD: No